CLINICAL TRIAL: NCT02164474
Title: Time-efficient High-intensity Interval Training Versus Moderate-intensity Continuous Aerobic Training for Promoting Exercise Adherence: A Randomized-controlled Trial
Brief Title: Small Steps for Big Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H12-02268
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Intensity Interval Training (HIIT) (Experimental): Participants will perform a series of high-intensity intervals with an interval length of 60-seconds at 90% of peak aerobic capacity workload, and a rest length of 60-seconds.
  Interventions: Behavioral: High-Intensity Interval Training
- Moderate-Intensity Continuous Exercise (Active Comparator): Participants will engage in exercise at 45% of peak aerobic capacity workload.
  Interventions: Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Specifically, individuals randomized to HIIT will begin the intervention with four intervals lasting 1-minute each at ~85-90% peak oxygen uptake [VO2peak] and increasing to 10 X 1-min intervals by day 10 of the intervention. Individuals randomized to moderate-intensity exercise condition will begin the intervention with 20 minutes of continuous activity at ~55-60% V02peak and gradually increase the duration to 50 minutes by day 10 of the intervention.

SUMMARY:
Exercise is a proven strategy for preventing type 2 diabetes. Traditionally individuals have been prescribed moderate-intensity continuous aerobic exercise but adherence to this standard exercise program is dismal. High-intensity interval training (HIIT) is a novel form of exercise that involves brief, repeated bursts of vigorous exercise separated by periods of recovery. HIIT elicits many favourable cardiometabolic adaptations that are similar to traditional exercise but does so with a lower amount of exercise and in substantially less time than moderate-intensity continuous exercise. Therefore, HIIT has been touted as a "time-efficient" exercise strategy for improving health. Whether overweight individuals at risk for pre diabetes will show greater adherence to HIIT than moderate-intensity continuous exercise over the long-term (12-months) has not been tested. Because exercise adherence requires complex self-regulation, interventions designed to improve adherence should include a behavioural component. The investigators will assess adherence to HIIT and moderate-intensity continuous exercise over 12 months following a short-term (2 week) intervention of either HIIT or moderate-intensity continuous exercise. Both conditions will include a self-regulatory component targeted to increase participants' confidence to engage in regular, independent exercise. The results will help determine whether HIIT is a more feasible option for promoting exercise adherence for pre diabetes prevention than the traditional moderate-intensity continuous exercise. The investigators hypothesize that a) over the 12 months follow-up subjects randomized to the HIIT will be more likely to adhere when compared to moderate-intensity continuous exercise, b) over the 12 months follow-up subjects randomized to HIIT will have higher rates of adherence and levels of total physical activity, c) greater increases in self-regulation (including goal setting, self-monitoring, and self-regulatory efficacy) following HIIT will mediate higher rates of adherence, d) 10-days of HIIT and moderate-intensity continuous exercise will improve cardiorespiratory fitness, increase insulin sensitivity, reduce circulating inflammatory markers, and improve glucose control and e) Improvements in cardiometabolic health factors will be greater following HIIT compared to moderate-intensity continuous exercise.

DETAILED DESCRIPTION:
Eligible participants will be randomized to the HIIT or moderate-intensity continuous exercise conditions. Each condition will involve a two-week supervised exercise period consisting of ten sessions. Exercise prescriptions for each condition will be progressive in nature over the two week supervised period and will be matched for external work. Specifically, individuals randomized to HIIT will begin with four intervals lasting 1-minute each at ~85-90% peak oxygen uptake [VO2peak] and increased to 10 X 1-min intervals by day 10. Individuals randomized to moderate-intensity exercise condition will begin with 20 minutes of continuous activity at ~55-60% V02peak and gradually increase the duration to 50 minutes by day 10. Participants will self-select exercise modality (walking outdoors, elliptical machine, treadmill walking, or stationary cycling). One trainer will supervise participants during the 2-week training program. Participants will complete 3 of the 10 training days (day 4, 7 and 9) at home unsupervised. Participants will wear a heart rate monitor during each exercise session (supervised and unsupervised) to monitor exercise intensity and ensure compliance. In addition, participants will record their exercise bouts in a logbook on both lab and home training days.

Participants in both conditions received 10 minutes of behavioural counseling each day they trained in the lab (for a total of 70 minutes). Following the supervised training, participants will be instructed to maintain HIIT or moderate-intensity continuous exercise three days per week independently. Specifically, individuals randomized to HIIT will be prescribed three exercise sessions per week involving 10 X 1-minute intervals at ~85-90% VO2peak, while participants randomized to moderate-intensity continuous exercise will be prescribed three session per week of 50-minute continuous exercise at ~55-60% VO2peak. Training logs will be provided and participants will be instructed to estimate exercise intensity based on physiological cues taught during supervised training days.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-65
* Physically inactive (engaging in 2 or less aerobic exercise bouts per week in the last 6 months)
* BMI between 24-40 kg/m2
* Cleared to engage in vigorous exercise (via PARQ+ and, if advised by this validated tool further clearance by their family physician)

Exclusion Criteria:

* Any contraindications to exercise (e.g., musculoskeletal injury)
* Failure to obtain medical clearance to engage in vigorous intensity exercise following a positive PARQ+ screening
* Prior history of cardio- or cerebrovascular disease or myocardial infarction
* Diagnosed with type 2 diabetes
* Currently taking glucose-lowering medications (e.g., metformin), Hypertension that is not controlled by medication (systolic blood pressure (BP) >160 mmHg and/or diastolic BP >99 mmHg)
* Change in cardiovascular medications (e.g., statins) in the previous 6 months Class III obesity (BMI >40 kg/m2).

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cardiorespiratory fitness (VO2peak) at 6 and 12-month follow-up | Baseline, 6-month follow-up and 12-month follow-up
  Changes in cardiorespiratory fitness (VO2peak), an objective measure of fitness and habitual activity, will be used as an integrative measure of exercise adherence (and overall health) at 6-month and 12-month follow-up. Specifically, peak oxygen uptake (VO2peak) will be assessed by a maximal cycling exercise test. Power output will begin at 30 W and increase by 15 W/min until volitional exhaustion. Expired gas samples will be collected continuously and VO2 measured by a metabolic cart (Parvomedics TrueOne 2400). The mean of the two highest 30 s average values will define VO2peak. VO2peak will be confirmed using standard criteria110. A Polar chest strap, which is integrated to the metabolic cart and cycle ergometer (Lode Excalibur), will capture Heart Rate. Peak power output will be recorded as the highest value attained.

SECONDARY OUTCOMES:
Self reported adherence to exercise prescription | Exercise log book filled in for a 12-month duration
  Self-reported adherence will be measuring using an online exercise log book, which participants will be asked to fill in following each exercise session. Adherence will be measured using raw exercise prescription bouts completed. Proportion achieved based on the amount prescription will also be calculated.
Changes from baseline in objectively measured moderate-to-vigorous physical activity in bouts ≥10 minutes (MVPA10+) at 3-, 6-, 9-, and 12-months follow-up | Baseline, 3-, 6-, 9-, 12-month follow-up
  Changes in total time spent in moderate-to-vigorous physical activity in bouts ≥10 minutes (MVPA10+) will be assessed over 7 days using tri-axial accelerometers at baseline and 3, 6-, 9- and 12-month follow-up.
Changes in efficacy beliefs | Baseline, Post-Intervention, 6-, 12-month follow-up
  Changes in participants exercise efficacy beliefs, self-regulatory efficacy beliefs, concurrent self-regulatory efficacy beliefs, and self-monitoring efficacy beliefs will be measured at baseline, post-intervention, 6-month follow-up and 12-month follow-up. Efficacy measures will be context specific and will utilize a confidence scale ranging from 0%-100%.
Changes in body composition | Baseline, post Intervention, 12-month follow-up
  Body composition will be assessed using the Hologic Discovery A device. DXA is a standard tool in the measurement of body composition and bone density in adults and children throughout multiple institutions.

OTHER OUTCOMES:
Changes in insulin sensitivity and inflammation | Baseline, post-intervention, 12-month follow-up
  Changes in insulin sensitivity and inflammation will be examined. Specifically fasting blooding samples will be taken to assess markers of insulin sensitivity (glucose, insulin, HOMA-IR) and inflammation (C-reactive protein [CRP], interleukin [IL]-6, tumor necrosis factor [TNF]-alpha).
Changes in acute affect during exercise sessions | Repeated measurements on Day 1, Day 6 and Day 9 of the intervention
  The acute affective response to exercise will be assessed using the 1-item Feeling Scale (FS). The FS is the most frequently used measure of in-task exercise feelings of pleasure/displeasure. Consistent with our established laboratory protocol for assessing and comparing affect in intermittent and continuous exercise bouts, feeling scale will be assessed immediately pre- and post-exercise, and at the beginning (2.5%), middle (42.5%), and end (92.5%) of workout completion. These time points correspond to the midpoint of the first, fifth, and tenth interval within the HIIT protocol. Measurements of affect will be taken in Day 1, Day 6 and Day 9 of the 10-day intervention.
Changes in exercise enjoyment | Baseline, post intervention, 6- and 12-month follow-up
  The Physical Activity Enjoyment Scale (PACES) will be used to assess perceived enjoyment at baseline and post intervention. This 18-item measure is scored on a 7-point bipolar scale based on the instruction; "Please rate how you feel at the moment about the physical activity you have been doing:". Example items are "it's not very refreshing/It's very refreshing" and "I would rather be doing something else/there is nothing else I would rather be doing". Items are summed to produce an overall enjoyment score out of 126.
Changes from baseline in average blood glucose at day 9 of the intervention | Baseline, Intervention day 9
  Changes in average blood glucose from baseline to day 9 of the intervention will be measured using the CGMS iPro2 (Medtronic, Northridge, CA). The CGM records glucose values in a blinded fashion using a small microneedle inserted into the subcutaneous abdominal adipose tissue that is connected to a recorder that quantifies interstitial glucose values every 5 minutes for up to three days. Finger stick blood glucose samples, taken four times per day, are used as calibrators to create a 24-hr blood glucose curve, which are downloaded upon device removal and analyzed for: i) average blood glucose, ii) 2 hr postprandial area under the glucose curve, iii) post-meal spikes, and iv) overall glycemic stability. Participants wearing the CGM will be provided a standardized diet (~24 kcal/kg, 60% carbohydrates, 27% fat, 13% protein) to consume during each 24 hr monitoring period. CGM data will be collected at baseline and day 9 of training.
Change in Affective and Instrumental Attitudes | Baseline, intervention day 6, post-intervention, 12-month follow-up
  Affective attitudes towards physical activity will be assessed using the procedures outlined by Ajzen (2002). Specifically, a 7-point semantic differential scale will be used, with anchors including "Enjoyable-Unenjoyable", "Pleasant-Unpleasant", "Interesting-Boring". Previous research has found support for both the internal consistency and predictive utility of scores derived from this instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Jung, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Health and Exercise Psychology Laboratory, Kelowna, British Columbia, Canada

REFERENCES:
- [Background] Little JP, Safdar A, Wilkin GP, Tarnopolsky MA, Gibala MJ. A practical model of low-volume high-intensity interval training induces mitochondrial biogenesis in human skeletal muscle: potential mechanisms. J Physiol. 2010 Mar 15;588(Pt 6):1011-22. doi: 10.1113/jphysiol.2009.181743. Epub 2010 Jan 25. PMID 20100740
- [Background] Little JP, Gillen JB, Percival ME, Safdar A, Tarnopolsky MA, Punthakee Z, Jung ME, Gibala MJ. Low-volume high-intensity interval training reduces hyperglycemia and increases muscle mitochondrial capacity in patients with type 2 diabetes. J Appl Physiol (1985). 2011 Dec;111(6):1554-60. doi: 10.1152/japplphysiol.00921.2011. Epub 2011 Aug 25. PMID 21868679
- [Background] Hood MS, Little JP, Tarnopolsky MA, Myslik F, Gibala MJ. Low-volume interval training improves muscle oxidative capacity in sedentary adults. Med Sci Sports Exerc. 2011 Oct;43(10):1849-56. doi: 10.1249/MSS.0b013e3182199834. PMID 21448086
- [Background] Trost SG, Owen N, Bauman AE, Sallis JF, Brown W. Correlates of adults' participation in physical activity: review and update. Med Sci Sports Exerc. 2002 Dec;34(12):1996-2001. doi: 10.1097/00005768-200212000-00020. PMID 12471307
- [Background] Jung ME, Wright WL, Wright AE, Ainslie PN, Little JP. Does the Relationship Between Affect and Exercise Intensity Apply to High-Intensity Interval Exercise? Medicine & Science in Sports & Exercise. 2012;44(5S):85.
- [Derived] Bourne JE, Little JP, Beauchamp MR, Barry J, Singer J, Jung ME. Brief Exercise Counseling and High-Intensity Interval Training on Physical Activity Adherence and Cardiometabolic Health in Individuals at Risk of Type 2 Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Mar 26;8(3):e11226. doi: 10.2196/11226. PMID 30912761
- [Derived] Bourne JE, Ivanova E, Gainforth HL, Jung ME. Mapping behavior change techniques to characterize a social cognitive theory informed physical activity intervention for adults at risk of type 2 diabetes mellitus. Transl Behav Med. 2020 Aug 7;10(3):705-715. doi: 10.1093/tbm/ibz008. PMID 30715534
- [Derived] Barry JC, Simtchouk S, Durrer C, Jung ME, Mui AL, Little JP. Short-term exercise training reduces anti-inflammatory action of interleukin-10 in adults with obesity. Cytokine. 2018 Nov;111:460-469. doi: 10.1016/j.cyto.2018.05.035. Epub 2018 Jun 6. PMID 29885989